CLINICAL TRIAL: NCT05379257
Title: A Feasibility Non-inferiority Clinical Trial for Dosing of Diuretics in CHF Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hadassah Medical Organization (Other)
Responsible Party: Principal Investigator, Dean Nahman, Physician, Hadassah Medical Organization
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RANDFURO- HMO-CTIL
Record Dates: First submitted 2020-12-06; First posted 2022-05-18 (Actual); Last update posted 2022-05-18 (Actual); Status verified 2022-05

CONDITIONS: Congestive Heart Failure
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Random dose (Experimental): Random dosage and timing of furosemide
  Interventions: Combination Product: Random dosage and time of furosemide

INTERVENTIONS:
Combination Product: Random dosage and time of furosemide — Random dosage and time of furosemide, using a designated app

SUMMARY:
Patients with heart failure are frequently hospitalized, have a reduced quality of life and face a higher risk of death. Much of the morbidity and reduced quality of life associated with CHF is related to symptoms of volume overload. Loop diuretics are a mainstay in the management of volume overload and edema in CHF.

Diuretic resistance is defined as the clinical state in which diuretic response is diminished or lost before the goal of treatment has been achieved. Diuretic resistance has an adverse effect on clinical outcomes and is associated with a poor prognosis.

This open-labeled study will evaluate the option to overcome this resistance in patients with partial of complete loss of the effect via random drug administration using an app. In the present study, the investigators will add the use of a treatment schedule prepared by the physician for each of the patients. This schedule includes a treatment regimen based on the drugs the patient is taking in a pre-determined random change within their approved therapeutic window to be administered by an app.

Patients will be followed for 10 weeks and will be compared with their pre-intervention condition. The effect and safety of altering the treatment regimen will be assessed by the need for intravenous diuretics, hospitalizations and emergency department admission and by Kansas City Cardiomyopathy Questionnaire (KCCQ), 6 minutes walk test, creatinine level and pro BNP levels.

DETAILED DESCRIPTION:
The objective of this study is to show non-inferiority in dosing diuretics using an app compared with standard of care, and to determine the safety and efficacy of using a diuretic dosing regimen provided by an app when administered to CHF patients with diuretic resistance.

Following 4 weeks of stabilization where all patients participating in the trial will receive their diuretics dosing in the conventional way by their health care provider, ten patients will start a 10-week intervention where they will be taking diuretics according to an irregular schedule which is within a range that was determined by their physician and within the therapeutic window. The app will change the dose and time in the day of taking the diuretics within the pre-determined ranges.The physician is required to provide each patient with a dosing range for his diuretics, while keeping the therapy within the approved therapeutic window. Irregularity is made daily by the app. Each patient will serve as his or her own control by comparing the effect of using the app to the effects of diuretics administered over the four weeks' period when he was using the diuretics without an app.

Patients will be monitored for safety that will be evaluated with creatinine level (normal values 62-115micromol/L higher values represent worsen kidney function), decompensation as determined by number of ER visits requiring intravenous diuretics and hospitalizations, and heart failure status that will be evaluated by diuretics dosage. Efficacy will be evaluated with KCCQ score (possible range of 0-100 better score represents better functional status), NT-proBNP levels (normal values 0-125 pg/ml) and 6 minutes walking test.

ELIGIBILITY:
Inclusion Criteria:

Ages Eligible for Study: 18 Years to 80 Years (Adult) Sexes Eligible for Study: All

1. Patients with NYHA II-III HFrEF, mid-range HF and HFpEF according to ESC definitions.
2. Patients taking at least 80 mg of furosemide daily in the 60 days previous to enrollment.
3. Females of childbearing potential must be non-pregnant (as determined by a serum pregnancy test at screening and again, prior to each dosing session) and agree to use adequate contraceptive means throughout the study.
4. No history of drug or alcohol abuse.
5. Patients must be able to adhere to the visit schedule and protocol requirements and be available to complete the study.
6. Patients must satisfy a medical examiner about their fitness to participate in the study.
7. Patients must provide written informed consent to participate in the study.

Exclusion Criteria:

1. Patients with evidence of other serious infectious, malignant, autoimmune, kidney, hepatic, or other non-cardiac systemic disease.
2. A major change in chronic therapies within 4 weeks.
3. Over-the-counter drugs, including herbal medications, and prescription drugs (other than those listed above) are not allowed for 4 weeks prior to and throughout the duration of the study
4. Participation in another clinical trial within 30 days prior to intervention.
5. Patients with an inability to communicate well with the Principal investigator (PI) and staff (i.e., language problem, poor mental development or impaired cerebral function).
6. Patients who will be unavailable for the duration of the trial, are likely to be noncompliant with the protocol, or who are felt to be unsuitable by the PI for any other reason.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Estimated)
Dates: Start 2020-01-20 (Actual); Primary Completion 2022-12-01 (Estimated); Study Completion 2022-12-01 (Estimated)

PRIMARY OUTCOMES:
Safety outcome | 10 weeks
  Patients will be monitored for safety that will be evaluated with creatinine level (normal values 62-115micromol/L higher values represent worsen kidney function), decompensation as determined by number of ER visits requiring intravenous diuretics and hospitalizations and higher diuretic dosage as a presentation of worsen heart failure
Efficacy outcome | 10 weeks
  KCCQ (possible range of 0-100 better score represents better functional status), NT-proBNP levels (normal values 0-125 pg/ml), 6 minute walk test in which higher walking distance represents better outcome

CONTACTS AND LOCATIONS:
Locations (1):
- Hadassah Medical Organization, Jerusalem, Israel

IPD SHARING:
Plan to Share IPD: No